CLINICAL TRIAL: NCT05226884
Title: Intermediate Vision in Patients With Clareon IOLs Compared to Eyhance IOLs
Status: Completed | Type: Observational
Sponsor: Berkeley Eye Center (Other)
Responsible Party: Sponsor
Other Study IDs: 69901155
Record Dates: First submitted 2022-01-04; First posted 2022-02-07 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Pseudophakia
Keywords: Clareon; Eyhance; pseudophakia
MeSH Terms: conditions — Pseudophakia | interventions — Visual Acuity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Clareon IOL Group: Patients with bilateral implantation of Clareon IOLs.
  Interventions: Diagnostic Test: Visual Acuity; Diagnostic Test: Defocus Curve
- Eyhance IOL Group: Patients with bilateral implantation of EyhanceIOLs.
  Interventions: Diagnostic Test: Visual Acuity; Diagnostic Test: Defocus Curve

INTERVENTIONS:
Diagnostic Test: Visual Acuity — Measurement of distance and intermediate visual acuity at variety targeted correction.
Diagnostic Test: Defocus Curve — Measurement of a defocus curve

SUMMARY:
Compare visual outcomes in patients with bilateral Clareon Monofocal IOLs versus bilateral Eyhance IOLs.

DETAILED DESCRIPTION:
This is a non-interventional prospective, comparative study of the outcomes for patients following successful, uncomplicated cataract surgery. All patients will have had bilateral implantation of an Eyhance IOL (DIB00/DIU***) or Clareon IOL (CNA0T0) at the time of uncomplicated cataract surgery. These patients will then be assessed post-operatively to compare distance and intermediate visual acuities and a defocus curve in patients with bilateral Clareon Monofocal IOLs versus bilateral Eyhance IOLs.

Patients will be assessed for corrected binocular distance and intermediate vision.

ELIGIBILITY:
Inclusion Criteria:

1. Adults, 40 years of age having already undergone uncomplicated cataract removal by phacoemulsification with a clear corneal incision in both eyes.
2. Implantation of bilateral Clareon intraocular lenses or Eyhance intraocular lenses (DIB00/DIU***).
3. Able to comprehend and willing to sign informed consent and complete all required testing procedures
4. Best Corrected Distance Visual Acuity (BCDVA) projected to be 0.10 logMAR (Minimum Angle of Resolution) or better
5. Clear intraocular media
6. Minimum of two weeks post yttrium aluminum garnet laser capsulotomy to treat PCO

Exclusion Criteria:

1. Any corneal abnormality, other than regular corneal astigmatism (as determined by pre-operative testing) that in the opinion of the investigator would confound the outcome(s) of the study
2. Any complication during cataract surgery (capsular tear, vitrectomy, etc)
3. History of or current retinal conditions in either eye that would confound the results of this investigation in the opinion of the investigator (e.g. retinal detachment, epiretinal membrane, retinal ischemia, retinal inflammation, etc)
4. Amblyopia or strabismus in either eye
5. History of or current anterior or posterior segment inflammation of any etiology
6. Any form of neovascularization on or within the eye
7. Glaucoma (uncontrolled or controlled with medication)
8. Optic nerve atrophy
9. Subjects with diagnosed degenerative eye disorders
10. Postoperative CDVA worse than 0.10 logMAR (20/25 snellen) in either eye.
11. Subjects who have an acute or chronic disease or illness that would confound the results of this investigation in the opinion of the investigator (e.g. immunocompromised, connective tissue disease, clinically significant atopic disease, etc)

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with healthy eyes and uncomplicated bilateral implantation of Eyhance intraocular lenses or Clareon intraocular lenses.
Sampling Method: Non-Probability Sample
Enrollment: 310 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-08-06 (Actual); Study Completion 2022-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Micheletti, MD, Principal Investigator — Berkeley Eye Center
Locations (1):
- Berkeley Eye Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Clareon IOL Group: Patients with bilateral implantation of Clareon IOLs who meet the inclusion/exclusion criteria.
  Visual Acuity: Measurement of distance and intermediate visual acuities
  Defocus Curve: Measurement of a defocus curve
  Refraction: Measurement of residual astigmatism and spherical equivalent.
- Eyhance IOL Group: Patients with bilateral implantation of Eyhance IOLs who meet the inclusion/exclusion criteria.
  Visual Acuity: Measurement of distance and intermediate visual acuities
  Defocus Curve: Measurement of a defocus curve
  Refraction: Measurement of residual astigmatism and spherical equivalent.
Period: Overall Study
Arm/Group | Clareon IOL Group | Eyhance IOL Group
Started | 155 | 155
Completed | 155 | 155
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clareon IOL Group | Eyhance IOL Group | Total
Number analyzed (Participants) | 155 | 155 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.26 (6.61) | 69.54 (6.85) | 69.45 (6.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 85 | 185
  Male | 55 | 70 | 125
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 6 | 3 | 9
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 52 | 16 | 68
  White | 94 | 134 | 228
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 155 | 155 | 310
Axial Length [Mean (Standard Deviation); unit: millimeters] — Axial length is obtained using an optical biometer prior to surgery and is a factor used to determine the power of the IOL to be implanted.
  millimeters | 23.81 (1.07) | 24.27 (1.41) | 24.04 (1.24)
IOL Power [Mean (Standard Deviation); unit: Diopters] — IOL power is determined using an optical biometer which takes various measurements of the eye to determine the lens power that should present the best visual outcome for the patient postoperatively.
  Diopters | 20.52 (2.86) | 19.77 (4.01) | 20.15 (3.44)
Corneal Astigmatism [Mean (Standard Deviation); unit: diopters] — Corneal astigmatism is the measure of the curvature of the cornea, which affects the way light is refracted which can cause a blurry image. Corneal astigmatism is measured during a refraction using a phoropter.
  diopters | 43.48 (1.49) | 43.08 (1.85) | 43.28 (1.67)
Anterior Chamber Depth [Mean (Standard Deviation); unit: millimeters] — Anterior chamber depth is obtained using an optical biometer prior to surgery and is a factor used to determine the power of the IOL to be implanted.
  millimeters | 3.13 (0.39) | 3.23 (0.39) | 3.18 (0.39)
Pupil Size [Mean (Standard Deviation); unit: millimeters] — Pupil size is obtained using an optical biometer prior to surgery and is a factor used to determine the power of the IOL to be implanted.
  millimeters | 3.61 (0.88) | 3.79 (0.86) | 3.7 (0.87)
Target/Aim [Mean (Standard Deviation); unit: diopters] — Diopter is a unit of measurement of the optical power of a lens, which is equal to the reciprocal of the focal length measured in meters.
  The target/aim is the goal for the visual outcome post-operatively. This may differ for each patient because it is based on lifestyle needs.
  diopters | -0.29 (0.32) | -0.29 (0.51) | -0.29 (0.42)
Predicted Post-operative Spherical Equivalent [Mean (Standard Deviation); unit: diopters] — Spherical equivalent is the estimate of each eye's refractive error. Predicted post-operative spherical equivalent is obtained using an optical biometer prior to surgery and is a factor used to determine the power of the IOL to be implanted.
  diopters | -0.32 (0.36) | -0.35 (0.52) | -0.34 (0.44)
Average Corneal Power [Mean (Standard Deviation); unit: Diopters] | 43.48 (1.49) | 43.01 (1.85) | 43.25 (1.67)

OUTCOME MEASURES:

1. Primary Outcome: Non-inferiority of Target-corrected Binocular Intermediate (66 cm) Visual Acuity With Offset
Description: Target-corrected binocular intermediate (66 cm) visual acuity of Clareon monofocal subjects at -0.25 sphere versus Eyhance subjects at plano sphere.
Time Frame: Minimum of 3 months post-operatively from cataract surgery, up to 2 years
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Clareon IOL Group | Eyhance IOL Group
Number analyzed (Participants) | 155 | 155
LogMAR | 0.20 (0.1) | 0.19 (0.11)
Statistical Analysis 1: Comparison: Clareon IOL Group vs Eyhance IOL Group; Test type: Non-Inferiority — Non-inferiority defined as within 0.1 LogMAR (1 line on Snellen Chart); p < 0.05, Wilcoxon (Mann-Whitney); Normality was assumed if skewness was ±2 and kurtosis was ±7. Non-inferiority was confirmed before further statistical testing

2. Primary Outcome: Non-inferiority of Distance Corrected Binocular Intermediate Visual Acuity
Description: Distance corrected binocular intermediate visual acuity (measured at 66 cm) of Clareon subjects versus Eyhance subjects with both groups set at plano sphere. Non-inferiority defined as 1 line.
Time Frame: Minimum of 3 months post-operatively from cataract surgery, up to 2 years
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Clareon IOL Group | Eyhance IOL Group
Number analyzed (Participants) | 155 | 155
LogMAR | 0.24 (0.11) | 0.19 (0.11)
Statistical Analysis 1: Comparison: Clareon IOL Group vs Eyhance IOL Group; Test type: Non-Inferiority — Non-inferiority defined as within 0.1 LogMAR (1 line on Snellen Chart); p < 0.05, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]

3. Primary Outcome: Non-inferiority of Best Corrected Distance Visual Acuity
Description: Comparison of Best Corrected Distance Visual Acuity (measured at 4m) of Clareon subjects versus Eyhance subjects.
Time Frame: Minimum of 3 months post-operatively from cataract surgery, up to 2 years
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Clareon IOL Group | Eyhance IOL Group
Number analyzed (Participants) | 155 | 155
LogMAR | 0.01 (0.02) | 0.02 (0.03)
Statistical Analysis 1: Comparison: Clareon IOL Group vs Eyhance IOL Group; Test type: Non-Inferiority — Non-inferiority defined as within 0.1 LogMAR (1 line on Snellen Chart); p < 0.05, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]

4. Primary Outcome: Binocular Distance Corrected Defocus Curve
Description: The Binocular Distance Corrected Defocus Curve measures visual acuity across simulated distances (+1.0D to -3.0D) in subjects with intraocular lenses (IOLs) post-cataract surgery. Testing begins with the best corrected visual acuity (BCVA), and the patient's refractive error is entered into the phoropter as the 0 position. Defocus lenses are introduced in 0.5D increments to simulate various distances. Visual acuity is measured binocularly at each level using standardized charts (e.g., ETDRS, Snellen) and recorded in logMAR. Measurements are taken at least 3 months post-op under standardized lighting conditions to evaluate visual performance across the defocus range in IOL patients.
Time Frame: Minimum of 3 months post-operatively from cataract surgery, up to 2 years
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Clareon IOL Group | Eyhance IOL Group
Number analyzed (Participants) | 155 | 155
LogMAR
  -3.0 D | 0.75 (0.17) | 0.74 (0.17)
  -2.5 D | 0.6 (0.17) | 0.58 (0.16)
  -2.0 D | 0.46 (0.16) | 0.44 (0.15)
  -1.5 D | 0.31 (0.13) | 0.29 (0.14)
  -1.0 D | 0.19 (0.11) | 0.16 (0.11)
  -0.5 D | 0.08 (0.07) | 0.07 (0.07)
  -0.25 D | 0.03 (.05) | 0.03 (.05)
  0 D | 0.01 (.02) | 0.02 (.03)
  0.25 D | 0.05 (.06) | 0.07 (0.07)
  0.5 D | 0.14 (.08) | 0.16 (.1)
  1 D | 0.31 (.12) | 0.31 (.11)
Statistical Analysis 1: Comparison: Clareon IOL Group vs Eyhance IOL Group; Test type: Non-Inferiority — Non-inferiority defined as within 0.1 LogMAR (1 line on Snellen Chart); The defocus curve is generated based on measurements over a dioptric range

5. Primary Outcome: Non-inferiority of Target-corrected Binocular Distance (4 m) Visual Acuity With Offset
Description: Target-corrected binocular distance (4 m) visual acuity of Clareon monofocal subjects at -0.25 sphere versus Eyhance subjects at plano sphere.
Time Frame: Minimum of 3 months post-operatively from cataract surgery, up to 2 years
Measure: Mean (Standard Deviation); unit: LogMAR
Arm/Group | Clareon IOL Group | Eyhance IOL Group
Number analyzed (Participants) | 155 | 155
LogMAR | 0.03 (0.02) | 0.02 (0.03)
Statistical Analysis 1: Comparison: Clareon IOL Group vs Eyhance IOL Group; Test type: Non-Inferiority — Non-inferiority defined as within 0.1 LogMAR (1 line on Snellen Chart); p < 0.05, Wilcoxon (Mann-Whitney); [statistical method as in outcome 1, analysis 1]

6. Secondary Outcome: Post-operative Spherical Equivalent
Description: Comparison of the Post-operative Spherical Equivalent of Clareon subjects versus Eyhance subjects.
Time Frame: Minimum of 3 months post-operatively from cataract surgery, up to 2 years
Measure: Mean (Standard Deviation); unit: Diopters
Arm/Group | Clareon IOL Group | Eyhance IOL Group
Number analyzed (Participants) | 155 | 155
Diopters | -0.04 (0.51) | -0.04 (0.73)

7. Secondary Outcome: Postoperative Residual Astigmatism
Description: Comparison of the amount of residual astigmatism of Clareon subjects versus Eyhance subjects.
Time Frame: Minimum of 3 months post-operatively from cataract surgery, up to 2 years
Measure: Mean (Standard Deviation); unit: Diopters
Arm/Group | Clareon IOL Group | Eyhance IOL Group
Number analyzed (Participants) | 155 | 155
Diopters | 0.43 (0.44) | 0.36 (0.36)

ADVERSE EVENTS:
Time Frame: Single (1 hour) visit
Description: Single visit, non-interventional study, meaning only visual acuity measurements were collected during a 1-hour study visit. All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were assessed but none were observed.
Arm/Group | Clareon IOL Group | Eyhance IOL Group
All-Cause Mortality (participants affected / at risk) | 0/155 | 0/155
Serious Adverse Events (participants affected / at risk) | 0/155 | 0/155
Other Adverse Events (participants affected / at risk) | 0/155 | 0/155

LIMITATIONS AND CAVEATS:
As this was a study on subjects who had already undergone cataract surgery, pre-operative targeting was not controlled for and based on patient discussions (e.g. mini-monovision, monovision, emmetropia). However, measuring visual acuities with distance correction allowed for a head-to-head comparison without residual postoperative refractive error as a confounding factor. Another potential limitation was that Eyhance torics were included, but the Clareon toric was not available.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-17): https://cdn.clinicaltrials.gov/large-docs/84/NCT05226884/Prot_SAP_000.pdf